CLINICAL TRIAL: NCT02909387
Title: Adapting Evidence-Based Epilepsy Self-Management Programs for Blacks in Georgia
Brief Title: Adapting Project UPLIFT for Blacks in Georgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Rakale Collins Quarells, Associate Professor, Morehouse School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GRANT11643642
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Epilepsy; Depressive Symptoms; Anxiety Disorders and Symptoms
Keywords: Epilepsy; Seizure Disorder
MeSH Terms: conditions — Epilepsy; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum A (Experimental): This group will be the first to receive the Project UPLIFT intervention, a distance-delivered mindfulness-based cognitive therapy intervention. The intervention is conducted by phone for one hour once a week for 8 weeks.
  Interventions: Behavioral: Project UPLIFT
- Stratum B (Active Comparator): This group will also receive the Project UPLIFT intervention at crossover, after a 10-week waiting period.
  Interventions: Behavioral: Project UPLIFT

INTERVENTIONS:
Behavioral: Project UPLIFT — UPLIFT is an 8-week distance-delivered mindfulness-based cognitive therapy intervention.
  Other Names: UPLIFT

SUMMARY:
Evaluate the efficacy of Project UPLIFT for reducing symptoms of depression and anxiety among African Americans at immediate posttest and after 3 months.

DETAILED DESCRIPTION:
Project UPLIFT is a manualized intervention that includes a script for use by the telephone facilitators in leading activities and discussions; use of a script is possible because the delivery is not face-to-face. Activities and discussions are designed to increase knowledge about epilepsy and mental health; monitoring, challenging, and changing of thoughts; coping and relaxing; attention and mindfulness; focusing on pleasure; the importance of reinforcement; and preventing relapse. Sessions are designed to last one hour by telephone, and are comprised of a check-in period, teaching on the topic of that week's session, group discussion, a skill-building exercise, and a recommended practice for the week. They are co-facilitated by a research staff and an UPLIFT trained adult with epilepsy. The same facilitators lead all eight sessions of a particular group. Facilitators will receive training in delivery of the program, including delivery of a practice session, from the Co-PI, a Georgia-licensed clinical psychologist. She will also supervise the facilitators throughout the program delivery. As noted above, spiritualism and religion; oral, interpersonal communication; and appreciation of intuition and experience are commonly held values in the African American community. This suggests that Project UPLIFT, with its activities based in experiential, meditative exercises, and oral, group discussion over the telephone may be a good fit.

Design. The outcome evaluation of the efficacy of the Project UPLIFT telephone intervention groups will be assessed using a cross-over design.

Participants/Procedure. A total of 60 participants will be recruited. Participants must self-identify as black or African American. All participants must be English-speaking, age 18 or older, mentally stable as assessed by the T-MMSE, have been diagnosed with epilepsy for at least three months, and screen positive for depression or anxiety on the Patient Health Questionnaire for Depression and Anxiety (PHQ-4). They must also have access to a telephone, be willing to attend eight hour-long telephone groups, and be willing to be audio-recorded. Individuals who are on antidepressant medication will not be excluded from this study, since CBT has been demonstrated to have a greater effect on relapse prevention than antidepressant medication. Once recruited, participants will be randomly assigned to one of two strata, each comprised of five 6-person groups. After each 12-participant cohort is recruited, they will be randomly assigned to Stratum 1 (intervention) or Stratum 2 (treatment-as-usual waitlist). During weeks 1-4, all participants will be pre-tested. During weeks 5-10, participants in Stratum 1 will receive Project UPLIFT, while participants in Stratum 2 are called weekly for a brief check-in. During weeks 11-14, all participants will receive interim testing. During weeks 15-22, participants in Stratum 2 will receive Project UPLIFT. During weeks 23-26, all participants will be post-tested. Five months after the completion of their final UPLIFT session, participants will be contacted for a follow-up assessment.

During the intervention in stratum 1, stratum 2 will serve as a control. In addition, the design allows a replication of the results in the initial intervention group (stratum 1) by the delayed intervention group (stratum 2). By the end of the intervention, all 10 6-person groups will have received the intervention.

Research Strategy Conferencing Methods. In order for the participants to communicate with one another as well as the facilitators, the telecommunicated group intervention sessions will use GoToMeeting. This conferencing method allows the moderator to not only record the call but also to screening participants waiting to join the call with the option to accept or reject those waiting, dismiss in-meeting participants, lock the meeting as well as dial out to participants. Use of this service is free of charge to MSM faculty.

Measures

Screening Measures will include the following:

Mental Stability will be assessed using the T-MMSE. The T-MMSE measures cognitive status, based on questions regarding orientation to time and place, recall, attention, naming, repetition, and a three-stage command. It was adapted from the Mini-Mental State Examination, takes about 5-10 minutes to administer, and has been shown to be a valid form of the assessment.

Symptoms of Anxiety or Depression will be assessed using the Patient Health Questionnaire-4 (PHQ-4).This is a very brief self-report instrument containing 2 depression items and 2 anxiety items. It is a compilation of the PHQ-2111 and the GAD-2.

Suicidal Intent or Planning will be assessed with the following items revised from the Youth Risk Behavior Survey to include only the past month: (1) During the past month, did you ever seriously consider attempting suicide? (2) During the past month, did you make a plan about how you would attempt suicide?

Evaluation Measures will include the following:

Acceptability will be assessed using the 8-item Client Satisfaction Questionnaire (CSQ-8), which has been demonstrated to correlate with number of psychotherapy sessions attended, and therapy outcome.

Cost and Health Outcomes will be assessed at baseline using the self-report survey instrument developed by Lairson and colleagues.

Effectiveness of the intervention will be assessed by comparing changes in knowledge, skills, and epilepsy self management from pretest to interim test to posttest across the strata. Changes in anxiety, depression, or PTSD symptom scores will also be evaluated using the methods described below.

Knowledge and Skills will be assessed using a measure in prior studies of Project UPLIFT.This instrument includes two sections, one for knowledge and one for skills. The knowledge items have true-false responses. The skills items have Likert-scaled response options measuring the value of each skill and the frequency of use of that skill.

Self management will be assessed using the latest version of the Epilepsy Self Management Scale (ESMS). The current version of this instrument includes 38-items and takes about 10 minutes to complete. IT includes subscales for Medication Management, Information Management, Safety Management, Seizure Management, and Lifestyle Management.

Depressive Symptoms will be assessed using two different measures. The mBDI, a modified form of the Beck Depression Inventory (BDI), will be used as one measure of depressive symptoms at pretest,interim, posttest, and follow-up. The mBDI is a measure of depression severity during the past 2 weeks. It contains the original 21 items of the BDI, but adds a positive response category for each item, such that the responses are scaled from 0 (positive) to 4 (severe). As a result, the mBDI is better at detecting differences in depression when depression scores are low. The 21-item BDI has also been shown to be valid for assessing depression among persons with epilepsy. Administration takes 5 to 10 minutes. The second measure of depressive symptoms will be the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 10-item instrument that closely follows diagnostic criteria for Major Depression as cited in the Diagnostic and Statistical Manual of Psychiatric Disorders. The PHQ-9 has been validated for diagnosing Major Depressive Disorder in primary care and in obstetric-gynecologic patients. The PHQ-9 can also be used to identify Major Depressive Disorder.

Symptoms of Anxiety will be assessed using two measures that are parallel to those used for depressive symptoms. Like the BDI, the Beck Anxiety Inventory (BAI) is another 21-item, self-report instrument, but it asks about the past week. Response choices range from 0 (not at all) to 3 (severe). As with the BDI, administration takes 5 to 10 minutes. The second anxiety measure will be the 7-item General Anxiety Disorder (GAD-7), a 7-item scale developed and validated within a primary care setting. The scale can also be completed by the patient.

Symptoms of Post-traumatic Stress Disorder (PTSD) will be assess using the PTSD-8. It is comprised of 4 Intrusive items, 2 Avoidance items, and 2 Hypervigilance items, for a total of 8 items. Item responses are on a 4-point Likert scale from 1 (not at all) to 4 (all the time). Likert-scale scoring permits measurement of symptom severity. This instrument has been tested across a range of diverse trauma samples including whiplash patients, rape victims, and disaster victims.

Evaluation. Process evaluation data will be obtained from the attendance records of each intervention session. Outcome evaluation measures will include changes in knowledge, skills, self-efficacy, and symptoms of depression, anxiety, and PTSD. Data from the pretest, interim test, and post-test will be entered by a Research Assistant, using SPSS. Changes in knowledge, skills, and mental health symptoms will be assessed using repeated measures multivariate analyses of variance (MANOVAs) across the variable of time (pretest, interim). Maintenance will be assessed comparing follow-up to pretest, and follow-up to immediate post (interim for stratum 1, post-test for stratum 2).

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American or Black;
* Diagnosed by a healthcare provider with epilepsy or seizure disorder at least 3 months ago;
* Is mildly to moderately depressed or mildly to moderately anxious as determined by the PHQ-4;
* Willing to be audio-recorded during UPLIFT sessions

Exclusion Criteria:

* Reports suicidal ideation within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Modified Beck Depression Inventory | Post intervention (8 weeks)
  Measure of depressive symptoms over previous two weeks.
Beck Anxiety Inventory | Post intervention (8 weeks)
  Measure of anxiety symptoms over previous week.

SECONDARY OUTCOMES:
Modified Beck Depression Inventory | 3-months Post Intervention
  Measure of depressive symptoms over previous two weeks.
Beck Anxiety Inventory | 3-months Post intervention
  Measure of anxiety symptoms over previous week.

CONTACTS AND LOCATIONS:
Overall Officials: Rakale C Quarells, PhD, Principal Investigator — Morehouse School of Medicine; Nancy Thompson, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared with the Managing Epilepsy Well Network (MEW) database.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by December 2019. Data will remain with the MEW Network database indefinitely.
Access Criteria: Access to data will be through the MEW Network database steering board.